CLINICAL TRIAL: NCT02561936
Title: A Phase 1, Open-label, Randomized, 2-panel, 4-way Crossover Study in Healthy Adult Subjects to Assess the Rilpivirine Relative Bioavailability Compared to the 25-mg Oral Tablet and the Food Effect Following Single Dose Administration of Oral Pediatric Formulation Candidates
Brief Title: Relative Bioavailability of Three Oral Formulations Candidates of Rilpivirine for Potential Pediatric Use Compared to Oral Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Sciences Ireland UC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR107783; TMC278IFD1008 (Other: Janssen Sciences Ireland UC); 2015-002511-14 (EudraCT Number)
Record Dates: First submitted 2015-08-21; First posted 2015-09-28 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
Keywords: Healthy; EUDRANT; Rilpivirine
MeSH Terms: interventions — Rilpivirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Panel 1: Group 1 (Experimental): Participants will receive Treatment A (25 milligram [mg] rilpivirine [RPV] formulated as the oral tablet under fed condition [standardized breakfast]) followed by Treatment D (25 mg RPV formulated as granules formulation G002 [10 g of 2.5 mg/g granules, dispersed in water] under fed [standardized breakfast]) followed by Treatment B (25 mg RPV formulated as dispersible tablet formulation G007 [10*2.5 mg tablets, dispersed in water] under fed condition) followed by Treatment C (25 mg RPV formulated as dispersible tablet formulation G009-01 [10*2.5 mg tablets, dispersed in water] under fed condition).
  Interventions: Drug: Rilpivirine Oral Tablet; Drug: Rilpivirine formulation G007; Drug: Rilpivirine formulation G009-01; Drug: Rilpivirine formulation G002; Dietary Supplement: Standardized Breakfast
- Panel 1: Group 2 (Experimental): Participants will receive treatment B followed by treatment A then treatment C followed by treatment D.
  Interventions: Drug: Rilpivirine Oral Tablet; Drug: Rilpivirine formulation G007; Drug: Rilpivirine formulation G009-01; Drug: Rilpivirine formulation G002; Dietary Supplement: Standardized Breakfast
- Panel 1: Group 3 (Experimental): Participants will receive treatment C followed by treatment B then treatment D followed by treatment A.
  Interventions: Drug: Rilpivirine Oral Tablet; Drug: Rilpivirine formulation G007; Drug: Rilpivirine formulation G009-01; Drug: Rilpivirine formulation G002; Dietary Supplement: Standardized Breakfast
- Panel 1: Group 4 (Experimental): Participants will receive treatment D followed by treatment C then treatment A followed by treatment B.
  Interventions: Drug: Rilpivirine Oral Tablet; Drug: Rilpivirine formulation G007; Drug: Rilpivirine formulation G009-01; Drug: Rilpivirine formulation G002; Dietary Supplement: Standardized Breakfast
- Panel 2: Group 1 (Experimental): Participants will receive Treatment E (25 mg RPV formulated as dispersible tablet formulation G007 or G009-01 or as granules formulation G002 [10*2.5 mg tablets or 10 g of 2.5 mg/g granules, dispersed in water] under fed [standardized breakfast] condition) followed by Treatment H (25 mg RPV formulated as dispersible tablet formulation G007 or G009-01 or as granules formulation G002 [10*2.5 mg tablets or 10 g of 2.5 mg/g granules, dispersed in water] under fed [yoghurt] condition) followed by Treatment F (25 mg RPV formulated as dispersible tablet formulation G007 or G009-01 or as granules formulation G002 [10*2.5 mg tablets or 10 g of 2.5 mg/g granules, dispersed in water] under fasted condition) followed by Treatment G (25 mg RPV formulated as dispersible tablet formulation G007 or G009-01 or as granules formulation G002 [10*2.5 mg tablets or 10 g of 2.5 mg/g granules, dispersed in water] under fed [standardized breakfast] condition).
  Interventions: Drug: Rilpivirine formulation G007; Drug: Rilpivirine formulation G009-01; Drug: Rilpivirine formulation G002; Dietary Supplement: Standardized Breakfast
- Panel 2: Group 2 (Experimental): Participants will receive Treatment F followed by Treatment E then Treatment G followed by Treatment H.
  Interventions: Drug: Rilpivirine formulation G007; Drug: Rilpivirine formulation G009-01; Drug: Rilpivirine formulation G002; Dietary Supplement: Standardized Breakfast
- Panel 2: Group 3 (Experimental): Participants will receive Treatment G followed by Treatment F then Treatment H followed by Treatment E.
  Interventions: Drug: Rilpivirine formulation G007; Drug: Rilpivirine formulation G009-01; Drug: Rilpivirine formulation G002; Dietary Supplement: Standardized Breakfast
- Panel 2: Group 4 (Experimental): Participants will receive Treatment H followed by Treatment G then Treatment E followed by Treatment F.
  Interventions: Drug: Rilpivirine formulation G007; Drug: Rilpivirine formulation G009-01; Drug: Rilpivirine formulation G002; Dietary Supplement: Standardized Breakfast

INTERVENTIONS:
Drug: Rilpivirine Oral Tablet — Rilpivirine formulated as 25 mg oral tablet.
  Other Names: Edurant
  Arms: Panel 1: Group 1; Panel 1: Group 2; Panel 1: Group 3; Panel 1: Group 4
Drug: Rilpivirine formulation G007 — Rilpivirine G007 formulation as 10*2.5 mg tablets.
Drug: Rilpivirine formulation G009-01 — Rilpivirine G009-01 formulation as 10*2.5 mg tablets.
Drug: Rilpivirine formulation G002 — Rilpivirine G002 formulation as 10 g of 2.5 milligram per gram (mg/gm) granules.
Dietary Supplement: Standardized Breakfast — It will consist of (or its equivalent) 4 slices of bread, 2 slices of ham and/or cheese, butter, fruit preserve and 1 or 2 cups (up to 480 milliliter [mL]) of decaffeinated coffee or decaffeinated tea with milk and/or sugar, if desired (containing approximately fat: 21 gram (gm), carbohydrates: 67 gm, proteins: 19 gm; calories 533 kilocalorie (kcal) [189 kcal from fat, 268 kcal from carbohydrates, and 76 kcal from proteins]).

SUMMARY:
The purpose of this study is to compare the rate and extent of absorption of rilpivirine in healthy adult participants following: 1) administration of a single dose of two different oral dispersible tablet formulation candidates and of an oral granules formulation with that following administration of a single dose of the 25-milligram (mg) oral tablet (EDURANT), after a standardized breakfast; 2) administration of a single dose of one selected oral formulation candidate (a dispersible tablet or granules) in different fed conditions (standardized breakfast or yoghurt) and in the fasted state and breakfast and 3) administration of a single dose of one selected oral formulation candidate (a dispersible tablet or granules) dispersed in water or in orange juice, in fed condition (standardized breakfast).

DETAILED DESCRIPTION:
This is a Phase 1, open-label, randomized, 2-panel, 4-way crossover study in healthy adult participants to assess the relative bioavailability of rilpivirine following single dose administration of oral pediatric formulation candidates (two dispersible tablet formulations and one granules formulation), compared to the commercially available 25-mg tablet (EDURANT) and to assess the effect of food and different food constituents on the oral bioavailability of rilpivirine following single dose administration of one selected formulation candidate. The study will consist of 2 panels: Panel 1 and Panel 2. In each panel, participants will be randomized to receive treatment A, B, C, D and E, F, G, H, respectively. Pharmacokinetic parameters will be evaluated primarily. Safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be willing and able to adhere to the prohibitions and restrictions specified in the protocol and study procedures
* Participant must be healthy on the basis of a medical evaluation that reveals the absence of any clinically significant abnormality and includes a physical examination, medical history, vital signs, electrocardiogram (ECG), and the results of blood biochemistry and hematology tests and a urinalysis performed at screening. If there are abnormalities, the participant may be included only if the Investigator judges the abnormalities or deviations from normal to be not clinically significant. This determination must be recorded in the participant's source documents and initialed by the Investigator
* Female participant must be either postmenopausal(amenorrhea for at least 2 years and a serum follicle-stimulating hormone [FSH] level greater than or equal to (>) 40 international units per liter (IU/L) [to be confirmed at screening for all postmenopausal women]), OR permanently sterilized (eg, bilateral tubal occlusion [which includes tubal ligation procedures as consistent with local regulations], total hysterectomy, bilateral salpingectomy, bilateral oophorectomy) or otherwise incapable of becoming pregnant, and have a negative serum pregnancy test at screening
* Male participants heterosexually active with a woman of childbearing potential must agree to use two effective contraceptive methods during the study and for at least 90 days after receiving the last dose of study drugs and male participants must agree not to donate sperm during the study and for at least 90 days after receiving the last dose of study drug
* Participants must be non-smoking for at least 3 months prior to Screening

Exclusion Criteria:

* Female participants who are breastfeeding at Screening
* Participants with a history of any illness that, in the opinion of the Investigator, might confound the results of the study or pose an additional risk in administering study drug to the participants or that could prevent, limit or confound the protocol specified assessments. This may include, but is not limited to, renal dysfunction, significant cardiac, vascular, pulmonary, gastrointestinal (such as significant diarrhea, gastric stasis, or constipation that in the Investigator's opinion could influence drug absorption or bioavailability), endocrine, neurologic, hematologic, rheumatologic, psychiatric, neoplastic, or metabolic disturbances
* Participants with current hepatitis B infection (confirmed by hepatitis B surface antigen [HBsAg]) or hepatitis C infection (confirmed by hepatitis C virus [HCV] antibody), or human immunodeficiency syndrome-1 (HIV-1 ) or HIV-2 infection
* Participants with a history of drug or alcohol abuse according to Diagnostic and Statistical Manual of Mental Disorders (5th edition) (DSM-V) criteria within 5 years before screening or positive test result(s) for alcohol and/or drugs of abuse (including barbiturates, opiates, cocaine, amphetamines, methadone, benzodiazepines, methamphetamine, tetrahydrocannabinol, phencyclidine, and tricyclic antidepressants) at Screening
* Participants with a history of clinically relevant skin disease such as, but not limited to, dermatitis, eczema, drug rash, psoriasis, food allergy, or urticaria

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2015-10; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Up to Hour 168
  The Cmax is the maximum observed plasma concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Time (AUC [0-last]) | Up to Hour 168
  The AUC (0-last) is the area under the plasma concentration-time curve from time zero to last quantifiable time.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) | Up to Hour 168
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z); wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.

SECONDARY OUTCOMES:
Time to Reach Maximum Observed Plasma Concentration (Tmax) | Up to Hour 168
  The Tmax is defined as time to reach maximum observed analyte concentration.
Elimination Rate Constant (Lambda[z]) | Up to Hour 168
  Lambda(z) is first-order elimination rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log-linear phase of the drug concentration-time curve.
Elimination Half-Life (t1/2) | Up to Hour 168
  The elimination half-life (t1/2) is the time measured for the plasma concentration to decrease by 1 half to its original concentration. It is associated with the terminal slope of the semi logarithmic drug concentration-time curve, and is calculated as 0.693/lambda(z).
Number of Participants with Adverse Events | From signing of the informed consent form up to 30 days after last dose of study drug (Day 1)
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Number of Participants with Taste Questionnaire Score | 15 minutes after study drug intake in each treatment period in both panels
  The first part of the taste questionnaire rates sweetness, bitterness and flavour as well as overall acceptability in a 4-point scale (grading from worse to best). In the second part of the taste questionnaire the overall taste is assessed using a 5-point visual hedonic scale (categorical 5 point assessment).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Sciences Ireland UC Clinical Trial, Study Director — Janssen Sciences Ireland UC
Locations (1):
- Antwerp, Belgium